CLINICAL TRIAL: NCT00003705
Title: Phase I Study of BMS-184476 in Patients With Advanced Malignancies
Brief Title: BMS-184476 in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: San Antonio Cancer Institute (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066813; UTHSC-9785011072; BMS-CA154-001; SACI-IDD-97-21; NCI-V98-1499
Record Dates: First submitted 1999-11-01; First posted 2004-03-15 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2007-08

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — 7-methylthiomethylpaclitaxel

INTERVENTIONS:
Drug: BMS-184476

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of BMS-184476 in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose, dose limiting toxicity, recommended phase II dose, and safety of BMS-184476 in patients with advanced solid tumors. II. Determine the pharmacokinetic profile of BMS-184476 and its metabolites in these patients. III. Determine preliminary evidence of antitumor activity of BMS-184476 in these patients.

OUTLINE: This is an open label, dose escalation study. Patients receive BMS-184476 IV over 1 hour. Treatment is repeated every 21 days in the absence of disease progression or unacceptable toxicity. In the second part of the study, patients receive BMS-184476 IV over 1 hour weekly. Cohorts of 3-6 patients are treated at escalating doses of BMS-184476. The maximum tolerated dose is defined as the dose at which fewer than 2 of 6 patients experience dose limiting toxicity. Patients are followed every 4 weeks until toxicity is resolved.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed advanced solid tumors refractory to conventional anticancer therapy, or for which no effective therapy exists Measurable or evaluable disease No active brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: Absolute neutrophil count at least 2,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL ALT and AST no greater than 2.5 times upper limit of normal (ULN) Renal: Creatinine less than 1.5 times ULN Cardiovascular: No uncontrolled or significant cardiovascular disease No myocardial infarction within past 6 months No congestive heart failure (with or without therapy) No history of atrial or ventricular arrhythmias No history of second or third degree heart block Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No serious uncontrolled medical disorder or active infection No known hypersensitivity to drugs containing Cremophor EL No concurrent neurologic toxicity No dementia or altered mental status

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior immunotherapy Chemotherapy: At least 4 weeks since prior chemotherapy (6 weeks since nitrosoureas, mitomycin, or carboplatin) Prior taxane therapy allowed No other concurrent chemotherapy Endocrine therapy: At least 1 week since prior steroid therapy No concurrent hormonal therapy Radiotherapy: At least 4 weeks since prior wide field radiotherapy (involving at least 30% of the bone marrow) No concurrent radiotherapy Surgery: Not specified Other: No other concurrent experimental anticancer medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-11

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Hidalgo, MD, PhD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (2):
- United States (2):
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - San Antonio Cancer Institute, San Antonio, Texas

REFERENCES:
- [Background] Plummer R, Ghielmini M, Calvert P, Voi M, Renard J, Gallant G, Gupta E, Calvert H, Sessa C. Phase I and pharmacokinetic study of the new taxane analog BMS-184476 given weekly in patients with advanced malignancies. Clin Cancer Res. 2002 Sep;8(9):2788-97. PMID 12231518
- [Result] Hidalgo M, Aylesworth C, Hammond LA, Britten CD, Weiss G, Stephenson J Jr, Schwartz G, Patnaik A, Smith L, Molpus K, Felton S, Gupta E, Ferrante KJ, Tortora A, Sonnichsen DS, Skillings J, Rowinsky EK. Phase I and pharmacokinetic study of BMS-184476, a taxane with greater potency and solubility than paclitaxel. J Clin Oncol. 2001 May 1;19(9):2493-503. doi: 10.1200/JCO.2001.19.9.2493. PMID 11331328